CLINICAL TRIAL: NCT03045107
Title: Intracorporeal or Extracorporeal Ileocolic Anastomosis After Laparoscopic Right Colectomy.
Brief Title: Intracorporeal or Extracorporeal Anastomosis After Laparoscopic Right Colectomy.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Prof. Mario Morino, Professor, University of Turin, Italy
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CS 863
Record Dates: First submitted 2017-02-03; First posted 2017-02-07 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Colon Cancer; Anastomosis
Keywords: right colon; laparoscopic right colectomy; intracorporeal anastomosis; extracorporeal anastomosis; hospital stay; quality of life; costs
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: A big dressing covering all incisions will be applied at the end of each operation in both arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intracorporeal ileocolic anastomosis (IIA) (Experimental): After complete right colon mobilization and ileocolic and right colic vessels ligation, the proximal transverse colon and the terminal ileum are transected and a side-to-side anastomosis is fashioned with a laparoscopic stapler.
  Interventions: Procedure: Laparoscopic right colectomy with intracorporeal ileocolic anastomosis (IIA)
- Extracorporeal ileocolic anastomosis (Active Comparator): After complete right colon mobilization and ileocolic and right colic vessels ligation, the terminal ileum, right colon, and proximal transverse colon are exteriorized for bowel division through a small midline skin incision in the upper abdomen. Then, a primary ileocolic side-to-side handsewn or mechanical anastomosis is fashioned extracorporeally.
  Interventions: Procedure: Laparoscopic right colectomy with extracorporeal ileocolic anastomosis (EIA)

INTERVENTIONS:
Procedure: Laparoscopic right colectomy with intracorporeal ileocolic anastomosis (IIA) — After complete right colon mobilization and ileocolic and right colic vessels ligation, the proximal transverse colon and the terminal ileum are transected with a laparoscopic EndoGIA TM stapler (Covidien Medtronic). The antimesenteric side of the stapled ends of the transverse colon and terminal ileum are approximated by a stay suture tied intracorporeally and then held by the assistant. An antimesenteric enterotomy and an antimesenteric colotomy are made about 10 cm distal to the stapled ends of the transverse colon and terminal ileum, respectively. A side-to-side anastomosis is fashioned with a laparoscopic EndoGIA TM stapler (Covidien Medtronic). The enterotomies are then closed by two layers of reabsorbable sutures tied intracorporeally. The specimen is delivered through a small Pfannenstiel or a median incision. A big dressing covering all incisions will be applied, similar to that used for the EIA group.
  Arms: Intracorporeal ileocolic anastomosis (IIA)
Procedure: Laparoscopic right colectomy with extracorporeal ileocolic anastomosis (EIA) — After complete right colon mobilization and ileocolic and right colic vessels ligation, the terminal ileum, right colon, and proximal transverse colon are exteriorized for bowel division through a small midline skin incision in the upper abdomen. A primary ileocolic side-to-side handsewn or mechanical (with GIA stapler - Covidien Medtronic) anastomosis is fashioned and the bowel returned to the abdominal cavity. After reinduction of pneumoperitoneum, the lack of twists of the ileocolic anastomosis is checked. A big dressing covering all incisions will be applied.
  Arms: Extracorporeal ileocolic anastomosis

SUMMARY:
During the last few years, the laparoscopic right colectomy with intracorporeal ileocolic anastomosis (IIA) has been proposed as an alternative to laparoscopic right colectomy with extracorporeal ileocolic anastomosis (EIA) for the treatment of right colon tumors. However, the level of evidence coming from the currently available literature is low, based on the results of a few small and heterogeneous retrospective non-randomized studies. A randomised controlled trial is warranted to challenge these two procedures. The aim of this randomized controlled trial is to assess the outcomes after IIA or EIA after laparoscopic right colectomy for right colon tumors.

DETAILED DESCRIPTION:
While there are no differences in oncologic principles (no touch technique, proximal vessel ligation, lymphadenectomy) between laparoscopic right colectomy with IIA and EIA, potential advantages of IIA are: (1) no need for extensive mobilization of the transverse colon to reach the abdominal wall; (2) performing the anastomosis away from the abdominal wall may lead to reduced rates of superficial site infection; (3) a shorter incision for the specimen extraction may be associated with clinical benefits such as less pain and lower rates of superficial site infections; (4) laparoscopic visualization during the creation of the IIA may reduce unrecognized twisting of the terminal ileum mesentery, and (5) the ability to remove the specimen through any type of incision, with subsequent reduced risks of incisional hernias in case of Pfannenstiel incision when compared to midline or off-midline incisions.

Some retrospective and heterogeneous studies comparing perioperative outcomes after laparoscopic right colectomy with EIA and IIA have been published in the last decade, reporting controversial results. Furthermore, the results of recent metanalyses are challenged by the heterogeneity and the poor quality of the published studies. Lastly, no comprehensive economic evaluation of the two procedures have been performed yet.

Consecutive patients with right colon tumors are included in a randomized controlled trial. This is a single Institution prospective randomized controlled trial comparing the outcomes in patients undergoing laparoscopic right colectomy with IIA or EIA for right colon neoplasm. Eligible patients will be randomly assigned in a 1:1 ratio to undergo either laparoscopic IA or EA according to a list of randomization numbers with treatment assignments. This list will be computer generated. An Internet application will allow central randomization.

Cost analysis will be based on the following costs: surgical instruments (including re-usable trocars and disposable tools), operative room, routine postoperative surgical care, diagnosis and treatment of postoperative complications. Operative room costs include healthcare personnel, medications, and structure costs. To calculate the cost of each postoperative complication, the following items will be assessed: laboratory and microbiology analysis; medical, technical, and diagnostic services; surgical and therapeutic interventions; medications; prolonged hospital stay, and outpatient clinic follow-up. The mean length of hospital stay of uncomplicated patients will be the basis to calculate the prolonged hospital stay in each patient with complication. In patients who will develop multiple complications, resources used to treat each complication will be recorded separately.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with a solitary benign or malignant neoplasm localized in the right colon
* Patients aged 18 years or older
* Patients who give written informed consent

Exclusion Criteria:

* acute intestinal obstruction
* colon perforation;
* liver and/or lung metastases;
* multiple primary colonic tumors;
* scheduled need for synchronous intra-abdominal surgery;
* preoperative evidence of invasion of adjacent structures, as assessed by CT or ultrasonography;
* previous ipsilateral colon surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2020-01-31 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay | 1 month

SECONDARY OUTCOMES:
Length of incisions | At the end of the operation
Intraoperative complications | intraoperatively
Number of lymph nodes harvested | 3 weeks
  evaluation of the number of lymph nodes in the specimen on pathology report
30-day postoperative morbidity according to the Clavien-Dindo classification | 1 month
First gas and stool passage | 1 week
Evaluation of postoperative pain (VAS) | 1 week
  measurement of VAS scores
Duration of intravenous analgesic therapy | 1 week
Narcotics use rate | from day 1 to day 5 after surgery
  percentage of patients requiring narcotics after surgery
Reoperation rate | 1 week
Hospital readmission | 90 days
  rate and causes of hospital readmission
In-hospital costs | 60 days
  Cost analysis will be based on the following costs: surgical instruments (including re-usable trocars and disposable tools), operative room, routine postoperative surgical care, diagnosis and treatment of postoperative complications. Operative room costs included healthcare personnel, medications, and structure costs. To calculate the cost of each postoperative complication, the following items will be assessed: laboratory and microbiology analysis; medical, technical, and diagnostic services; surgical and therapeutic interventions; medications; prolonged hospital stay, and outpatient clinic follow-up. The mean length of hospital stay of uncomplicated patients will be the basis to calculate the prolonged hospital stay in each patient with complication. In patients who will develop multiple complications, resources used to treat each complication will be recorded separately.
Rate of incisional hernias | postoperatively at 3 and 6 months
Quality of life | preoperatively, at 3 and 6 months after surgery
  the SF-12 questionnaire will assess quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Mario Morino, MD, Principal Investigator — University of Turin, Italy
Locations (1):
- Department of Surgical Sciences, University of Torino, AOU Città della Salute e della Scienza, Torino, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hellan M, Anderson C, Pigazzi A. Extracorporeal versus intracorporeal anastomosis for laparoscopic right hemicolectomy. JSLS. 2009 Jul-Sep;13(3):312-7. PMID 19793468
- [Result] Fabozzi M, Allieta R, Brachet Contul R, Grivon M, Millo P, Lale-Murix E, Nardi M Jr. Comparison of short- and medium-term results between laparoscopically assisted and totally laparoscopic right hemicolectomy: a case-control study. Surg Endosc. 2010 Sep;24(9):2085-91. doi: 10.1007/s00464-010-0902-8. Epub 2010 Feb 21. PMID 20174945
- [Result] Grams J, Tong W, Greenstein AJ, Salky B. Comparison of intracorporeal versus extracorporeal anastomosis in laparoscopic-assisted hemicolectomy. Surg Endosc. 2010 Aug;24(8):1886-91. doi: 10.1007/s00464-009-0865-9. Epub 2010 Jan 29. PMID 20112118
- [Result] Chaves JA, Idoate CP, Fons JB, Oliver MB, Rodriguez NP, Delgado AB, Lizoain JL. [A case-control study of extracorporeal versus intracorporeal anastomosis in patients subjected to right laparoscopic hemicolectomy]. Cir Esp. 2011 Jan;89(1):24-30. doi: 10.1016/j.ciresp.2010.10.003. Epub 2010 Dec 19. Spanish. PMID 21176829
- [Result] Roscio F, Bertoglio C, De Luca A, Frattini P, Scandroglio I. Totally laparoscopic versus laparoscopic assisted right colectomy for cancer. Int J Surg. 2012;10(6):290-5. doi: 10.1016/j.ijsu.2012.04.020. Epub 2012 May 4. PMID 22564829
- [Result] Scatizzi M, Kroning KC, Borrelli A, Andan G, Lenzi E, Feroci F. Extracorporeal versus intracorporeal anastomosis after laparoscopic right colectomy for cancer: a case-control study. World J Surg. 2010 Dec;34(12):2902-8. doi: 10.1007/s00268-010-0743-6. PMID 20703468
- [Result] Milone M, Elmore U, Di Salvo E, Delrio P, Bucci L, Ferulano GP, Napolitano C, Angiolini MR, Bracale U, Clemente M, D'ambra M, Luglio G, Musella M, Pace U, Rosati R, Milone F. Intracorporeal versus extracorporeal anastomosis. Results from a multicentre comparative study on 512 right-sided colorectal cancers. Surg Endosc. 2015 Aug;29(8):2314-20. doi: 10.1007/s00464-014-3950-7. Epub 2014 Nov 21. PMID 25414066
- [Result] Hanna MH, Hwang GS, Phelan MJ, Bui TL, Carmichael JC, Mills SD, Stamos MJ, Pigazzi A. Laparoscopic right hemicolectomy: short- and long-term outcomes of intracorporeal versus extracorporeal anastomosis. Surg Endosc. 2016 Sep;30(9):3933-42. doi: 10.1007/s00464-015-4704-x. Epub 2015 Dec 29. PMID 26715015
- [Result] van Oostendorp S, Elfrink A, Borstlap W, Schoonmade L, Sietses C, Meijerink J, Tuynman J. Intracorporeal versus extracorporeal anastomosis in right hemicolectomy: a systematic review and meta-analysis. Surg Endosc. 2017 Jan;31(1):64-77. doi: 10.1007/s00464-016-4982-y. Epub 2016 Jun 10. PMID 27287905
- [Derived] Seno E, Allaix ME, Ammirati CA, Bonino MA, Arezzo A, Mistrangelo M, Morino M. Intracorporeal or extracorporeal ileocolic anastomosis after laparoscopic right colectomy: cost analysis of the Torino trial. Surg Endosc. 2023 Jan;37(1):479-485. doi: 10.1007/s00464-022-09546-7. Epub 2022 Aug 23. PMID 35999317
- [Derived] Allaix ME, Degiuli M, Bonino MA, Arezzo A, Mistrangelo M, Passera R, Morino M. Intracorporeal or Extracorporeal Ileocolic Anastomosis After Laparoscopic Right Colectomy: A Double-blinded Randomized Controlled Trial. Ann Surg. 2019 Nov;270(5):762-767. doi: 10.1097/SLA.0000000000003519. PMID 31592811